CLINICAL TRIAL: NCT02874859
Title: Aflibercept Injection for Treatment of Diabetic Macular Edema
Brief Title: Intravitreal Aflibercept InjectiOn in Vitrectomized Eyes for Treatment of Diabetic Macular Edema
Acronym: MODEVA
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: RC-P0051
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Macular Edema
Keywords: DIABETIC RETINOPATHY; Intravitreal aflibercept
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This a non-interventional retrospective study on the efficiency and the tolerance of intravitreal injections of Aflibercept on vitrectomized eyes in the diabetic macular oedema

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is the leading cause of blindness among people of working age. Treatment of DME included blood pressure and glycemic control, grid laser, intravitreal injection of steroids (acetonide of triamcinolone, dexamethasone implant, fluocinolone implant) or anti-Vascular endothelial growth factor (VEGF) therapy (Bevacizumab, Ranibizumab, Aflibercept) (2015). The advent of anti-VEGF therapy has revolutionized the management of DME. Aflibercept, one of the drugs in this group has recently been approved in France. However, there is no report in the efficacy and tolerance of Aflibercept in vitrectomized eyes in the diabetic macular oedema . In this study, in order to prove the efficiency and tolerance of Aflibercept, data will be collected in a anonymous way in medical records of patients having received a treatment by Aflibercept in the past.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients aged between 19 and 90 years old
* Patients with the following characteristics at the beginning of the Aflibercept therapy :

HbA1c < 9% Diabetic macular oedema with the central affected Visual acuity between 1/20 and 5/40 (between 20 and 70 letters ETRS) Patients who had a vitrectomy over 3 months ago

* Patients who did not received an anti-VEGF treatment or any other treatment for their diabetic macular edema 3 months before the beginning of the injections

Exclusion Criteria:

* Patients who refused the collection of their data in medical records
* Patients with a macular ischemia of more than 1500µm diagnosed via an avascular central fluorescein angiography before the inclusion
* Patients with a recent cardiovascular incident (heart attack, stroke dating for less than 3 months before the inclusion)
* Pregnancy at the moment of inclusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic vitrectomised patients with macular edema, treated with Aflibercept in the past
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Estimation of visual acuity Early Treatment Diabetic Retinopathy Study (ETDRS) | 96 weeks
  Estimation of visual acuity after 96 weeks of treatment with Aflibercept

SECONDARY OUTCOMES:
Measure of the central macular thickness | 96 weeks
  Describe the evolution of the Central macular thickness during treatment
Quantification of number of Aflibercept injections received | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thi Ha Chau TRAN, PhD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (8):
- France (8):
  - Pr MILAZZO Solange, Amiens, Hauts-de-France
  - Tran Thi Ha Chau, Lomme, Hauts-de-France
  - Stéphanie BAILLIF, Nice, PACA
  - Dr DOMINGUEZ, Bordeaux
  - Pr KODJIKIAN, Lyon
  - Dr Franck BECQUET, Nantes
  - Dr UZZAN, Rouen
  - Bénédicte DUPAS, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran THC, Erginay A, Verdun S, Fourmaux E, Le Rouic JF, Uzzan J, Milazzo S, Baillif S, Kodjikian L. One-Year Outcome of Aflibercept Intravitreal Injection in Vitrectomized Eyes with Diabetic Macular Edema. Clin Ophthalmol. 2021 May 11;15:1971-1978. doi: 10.2147/OPTH.S304030. eCollection 2021. PMID 34007150